CLINICAL TRIAL: NCT05065788
Title: Impact of COVID-19 Pandemic and Related Lockdown on Eye Emergencies Accesses
Brief Title: Ophthalmological Emergencies and COVID-19 Pandemia
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Simone Donati, Associate Professor, Università degli Studi dell'Insubria
Other Study IDs: 02/2021 - COVID and EYE
Record Dates: First submitted 2021-09-30; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Trauma; Infections; Vision; Loss, Both Eyes
Keywords: ocular emergency; vision loss
MeSH Terms: conditions — Wounds and Injuries; Infections; Blindness; Vision Disorders | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2020 Lockdown period: Patients who access to Ophthalmological emergency service during lockdown period in 2020
  Interventions: Other: data collection
- 2019: Patients who access to Ophthalmological emergency service in 2019 definite periods
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
To analyze how the COVID 19 pandemia has affected the patient's accesses to the Ophthalmological Emergency Department of a tertiary referral center in northern Italy, during the lockdown period. We will collect data from different periods in 2020, in which the Italian Governement called the total lockdown to same periods of the 2019. The charts of all patients will be evaluated to analyze demographics and clinical data

DETAILED DESCRIPTION:
Since the end of 2019, an outbreak of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), originating in the Chinese city of Wuhan has spread rapidly worldwide causing thousands of deaths. Coronavirus disease (COVID-19) is supported by SARS-CoV-2 and represents the causative agent of a potentially fatal disease that is of great global public health concern. Italy has been the first European country recording an elevated number of infected forcing the Italian Government to call for total lockdown. The lockdown had the aim to limit the spread of infection through social distancing. The purpose of this study is to analyze how the pandemic has affected the patient's accesses to the Ophthalmological Emergency Department of a tertiary referral center in northern Italy, during the lockdown period. The charts of all patients that came to the Emergency Department during the lockdown period (February -May, 2020 and October - December 2020) will be retrospectively collected and compared with those in the same periods of 2019 .

All demographics and clinical data will be analyzed and compared to evaluate differences and type of accesses.

ELIGIBILITY:
Inclusion Criteria:

Access to emergency room in the definite periods Completed Patients Charts -

Exclusion Criteria:

Access to emergency room in other periods Demographics and clinical data not completed

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered for access to emergency ophthalmological room in the periods:
  2020 from February to May and from October to December 2019 from February to May and from October to December
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
number of patients | 1 year
  evaluation of number of accesses

SECONDARY OUTCOMES:
Type of pathologies | 1 year
  Classification according to type of pathologies that causes the access to Emergency Room

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Sette Laghi, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poyser A, Deol SS, Osman L, Kuht HJ, Sivagnanasithiyar T, Manrique R, Okafor LO, DeSilva I, Sharpe D, Savant V, Sarodia U, Sarvananthan N, Chaudhuri R, Banerjee S, Burns J, Thomas MG. Impact of COVID-19 pandemic and lockdown on eye emergencies. Eur J Ophthalmol. 2021 Nov;31(6):2894-2900. doi: 10.1177/1120672120974944. Epub 2020 Nov 19. PMID 33213198
- [Result] Ehlken C, von Medem C, Ludemann M, Kirsch AM, Roider JB. Patients' perspective on emergency treatment of ophthalmologic diseases during the first phase of SARS-CoV2 pandemic in a tertiary referral center in Germany - the COVID-DETOUR questionnaire study. BMC Ophthalmol. 2021 Aug 16;21(1):301. doi: 10.1186/s12886-021-02054-7. PMID 34399720
- [Result] Salvetat ML, Salati C, Busatto P, Zeppieri M. The impact of COVID-19 related national lockdown on ophthalmic emergency in Italy: A multicenter study. Eur J Ophthalmol. 2022 May;32(3):1782-1794. doi: 10.1177/11206721211028046. Epub 2021 Jul 3. PMID 34219482